# Template onderzoeksprotocol niet-WMO plichtige studie

| STUDIEGEGEVENS | | | |
|---|---|---|---|
| Titel van de studie | Time within the Acute Care Chain: how long have medical emergency department patients spent? | | |
| Acroniem van de studie | TA | CC studie | |
| Soort studie | | retrospectief onderzoek | |
| | $\boxtimes$ | prospectief onderzoek | |
| Versienummer protocol | 2.0 | | |
| Datum protocol | 17 | -08-2021 | |
| Opdrachtgever studie | Zu | yderland | |
| Leden onderzoeksteam | Ge | egevens | Rol |
| | 1 | Lieke Claassen, SEH-arts <sup>KNMG</sup> | Hoofdonderzoeker/Coördinerend |
| | | Zuyderland | onderzoeker |
| | 2 | Gideon Latten, SEH-arts <sup>KNMG</sup> | Onderzoeker |
| | | Zuyderland | |
| | 3 | Patricia Stassen, internist acute | Onderzoeker |
| | 4 | geneeskunde MUMC+ | |
| Lokale hoofdonderzoeker | | ! | T-1-f |
| Lokale noordonderzoeker | Emailadres: | | Telefoonnummer: 0645955271 |
| | | laassen@zuyderland.nl | |
| Contactpersoon studie | Emailadres: | | Telefoonnummer: 0645955271 |
| I.claassen@zuyderland.nl | | | |
| Dit onderzoek wordt uitgevoerd in het kader van een | | | |
| onderzoekslijn van Zuyderland | | | |
| promotieonderzoek | | | |
| universitaire studie | | | |
| HBO studie | | | |
| anders, namelijk: | | | |

| 1 |
|------------|
| 2 |
| 3 |
| <u>3</u> 4 |
| 4 |
| 5 |
| 5 |
| 5 |
| 5 |
| 6 |
| 6 |
| 8 |
| 8 |
| 8 |
| 8 |
| 9 |
| 10 |
| 11 |

## **SAMENVATTING**

Deze studie is onderdeel van een onderzoekslijn naar de acute zorgketen, waarmee het traject bedoeld wordt van start van symptomen/klachten tot en met behandeling op de spoedeisende hulp (SEH). Het huidige onderzoek legt de focus op de zogeheten gehele patient journey en de doorlooptijd van patiënten door de acute zorgketen heen.

Bij veel aandoeningen is de tijd die het kost om tot behandeling over te gaan van belang. Een voorbeeld is een acuut myocardinfarct. Binnen ziekenhuizen is er veel aandacht voor triage, de doorlooptijd (m.n. op de SEH) en het voorkomen van vertraging in de behandeling van patiënten. Over de periode voorafgaand aan het SEH-bezoek is echter minder bekend. Eerder stelden wij vast dat de mediane duur van klachten van patiënten op de SEH met een infectie 3 dagen is, waarbij een kwart van de patiënten reeds antibiotica gebruikt had en 40% reeds eerder de huisarts bezocht had.¹ Echter, voor andere aandoeningen is dit nog niet goed bekend. Tevens is de verdeling van tijd per 'station' ((verpleeg-)huisarts, ambulance, SEH) niet bekend, alsook niet wat er in iedere schakel gebeurt. Meer inzicht in de gehele acute zorgketen en de "journey" van patiënten is essentieel voor verdere optimalisatie van de zorg voor alle SEH-patiënten.

In de Houtskoolschets acute zorg gaat men uit van specifieke patiëntengroepen. Een patiënt komt echter meestal niet met een duidelijke diagnose (bijvoorbeeld CVA of ernstig trauma) de keten in. Daarnaast wordt in de Houtskoolschets aangegeven dat de drukte op de SEH's toeneemt, het acute zorglandschap verandert en dat de zorg wellicht slimmer kan. Om dit te verbeteren moeten we wel weten hoe het huidige traject er uit ziet, juist voor de patiënten die niet meteen een duidelijke diagnose hebben. Tot voor kort was niet bekend hoe het traject van deze patiënten in de acute zorgketen eruit zag. Een pilotstudie binnen het Zuyderland MC liet zien dat een beschouwende patiënt gemiddeld 6 uur in de acute zorgketen doorbrengt en hierbij meerdere stations van zorgverleners passeert (METC nr Z2020228). Echter, dit betrof een pilot studie en niet de gehele patiëntenpopulatie op de Spoed Eisende Hulp. In het huidige onderzoek beogen wij in een grotere studie en regio breed de patient journey in de acute zorgketen te achterhalen.

In het huidige onderzoek zullen wij 750 patiënten includeren op diverse SEH's in de provincie Limburg. Te weten: Venlo, Weert, Roermond, Heerlen, Sittard-Geleen en Maastricht.

Het doel van het onderzoek is inzicht te krijgen in de routing van de acute patiënt, de doorlooptijd van de patiënt die de SEH bereikt, wat gebeurt er per station en wat is de uitkomst na de SEH?

De vragen die we met deze studie hopen te beantwoorden zijn als volgt:

 Primaire onderzoeksvraag: Hoe ziet de patient journey eruit van volwassen patiënten die met een acute zorgvraag de SEH bereiken?

Secundaire onderzoeksvragen:

- Wat is de doorlooptijd binnen de acute zorgketen van acuut zieke volwassen patiënten die met een acute zorgvraag de SEH bereiken?
- Hoe vaak heeft een patiënt contact gehad met een hulpverlener alvorens de SEH te bezoeken? Welke hulpverleners waren dit en met welk urgentieniveau?
- Wat gebeurt er in de tijd dat de patiënt zich in de acute zorgketen bevindt? Welke onderzoeken worden er gedaan?
- Wat gebeurt er nadat de patiënt op de SEH is geweest? Wat is de uitkomst van de patiënt die op de SEH is behandeld: opname reguliere afdeling, opname op bewaakte afdeling (IC/MC), mortaliteit binnen 7 en 30 dagen, herbezoek?

## 1. INTRODUCTIE

De spoedeisende hulp (SEH) is doorgaans de toegangspoort naar het ziekenhuis voor patiënten met een acute zorgvraag. Bij veel acute aandoeningen is de tijd die het kost om tot behandeling over te gaan van belang. Dit geldt niet alleen voor de 'bekende' acute aandoeningen zoals een traumatisch letsel, een hartinfarct, of een beroerte, maar ook voor aandoeningen als een infectie, een elektrolytstoornis, of een anemie. Echter, tijdens het eerste contact is vaak nog niet altijd duidelijk van welk ziektebeeld er sprake is.

De hoeveelheid van acute zorgcontacten en de drukte op de SEH's neemt toe en het zorglandschap is aan veranderingen onderhevig. In de Houtskoolschets acute zorg wordt aangegeven het acute zorglandschap te vernieuwen en te verbeteren ten aanzien van spoedposten, spoedeisende hulpen etc.. Echter, de schets focust op patiënten met duidelijke problemen als een acuut myocardinfarct, herseninfarct, vaatpathologie of traumatologie welke slechts minder dan de helft van de zorgstroom uitmaken.² Daar de patiënten populatie op de SEH meer omvat dan gedifferentieerde patiënten, lijkt de huidige stand van zaken onvoldoende in kaart is-gebracht. Inzicht in de gehele patiëntenstroom en de patient journey binnen de acute zorgketen van deze patiëntengroep kan bijdragen aan een oplossing voor dit landelijke

vraagstuk. Met de patient journey wordt de reis bedoeld van start van symptomen/klachten tot en met behandeling op de SEH.

Binnen ziekenhuizen is er veel aandacht voor triage, doorlooptijd (m.n. op de SEH) en het voorkomen van vertraging in de behandeling van patiënten met een acute zorgvraag. Echter, het merendeel van de bovengenoemde patiënten meldt zich niet primair op de SEH, maar bij de huisarts of ambulance dienst.<sup>1, 3</sup> Voor de meeste aandoeningen is niet bekend hoe patiënten door de acute zorgketen heen 'reizen', wat de doorlooptijd is in de gehele acute zorgketen, hoeveel zorgverleners patiënten al gezien hebben en wat er gebeurt binnen de diverse schakels ((verpleeg-)huisarts, ambulance, SEH) van de acute zorgketen.

Voor patiënten met een infectie zochten wij eerder uit hoe de prehospitale fase eruit ziet.¹ Deze patiënten hadden mediaan 3 dagen klachten, 40% had al eerder de huisarts bezocht en 25% gebruikte al antibiotica. Op de dag van het SEH bezoek was 80% van de patiënten verwezen door een huisarts. Deze data zijn niet bekend voor de meeste andere patiënten die niet direct in een diagnosecluster te plaatsen zijn en die buiten de Houtskoolschets vallen. In een eerdere pilot studie binnen Zuyderland zagen we dat een patiënt zich gemiddeld 6 uur in de acute zorgketen bevindt en hierbij meerdere stations van zorgverleners passeert. Echter, dit betrof een relatief kleine, single center pilot studie (METC NR Z2020228). In de huidige studie is het doel in een grotere, regio brede studie te achterhalen hoe de patient journey in de acute zorgketen eruit ziet van alle volwassen patiënten die met een acute zorgvraag op de SEH behandeld worden. Inzicht in de 'patient journey' binnen de acute zorgketen is onontbeerlijk voor de verder optimalisatie en verbetering van de om de acute zorgketen.

Deze studie is onderdeel van een onderzoekslijn naar de acute zorgketen, waarmee het traject bedoeld wordt van start van symptomen/klachten tot en met behandeling op de spoedeisende hulp (SEH). Het huidige onderzoek legt de focus op de gehele patiënt journey van acute zieke volwassen die op de SEH behandeld worden.

## 1.1 Onderzoeksvraag, - hypothese en/of -doel

De vragen die we met deze studie hopen te beantwoorden zijn als volgt:

 Primaire onderzoeksvraag: Hoe ziet de patient journey eruit van volwassen patiënten die met een acute zorgvraag de SEH bereiken?

Secundaire onderzoeksvragen:

- Wat is de doorlooptijd binnen de acute zorgketen van acuut zieke volwassen patiënten die met een acute zorgvraag de SEH bereiken?
- Hoe vaak heeft de patiënt contact gehad met een hulpverlener alvorens de SEH te bezoeken? Welke hulpverleners waren dit en met welk urgentieniveau?
- Wat gebeurt er in de tijd dat de patiënt zich in de acute zorgketen bevindt? Welke onderzoeken worden er gedaan?
- Wat gebeurt er nadat de patiënt op de SEH is geweest? Wat is de uitkomst van de patiënt die op de SEH is behandeld: opname reguliere afdeling, opname op bewaakte afdeling (IC/MC), mortaliteit binnen 7 en 30 dagen, herbezoek?

## 2. METHODEN

## 2.1 Studieprocedure/study design

Dit is een prospectieve multicenter observationele studie. De studie vindt tegelijkertijd plaats op alle SEH's in Limburg, te weten: Maastricht, Heerlen, Sittard, Roermond, Weert en Venlo. De studie zal plaatsvinden volgens de flashmobmethode waarmee in een kort tijdsbestek van 72 uur ongeveer 750 patiënten geïncludeerd zullen worden.<sup>4</sup>

## 2.2 Werving en selectie van proefpersonen

## Studiepopulatie

Alle patiënten van 18 jaar of ouder die behandeld worden op een SEH in Limburg zullen geïncludeerd worden. Alle patiënten wordt informed consent gevraagd.

## Screening/selectie

Patiënten worden gescreend en geïncludeerd door een student, een arts klinisch onderzoeker (AKO) i.o., een A(N)IOS, een SEH-arts<sup>KNMG</sup> of een medisch specialist. In principe komen alle patiënten die voldoen aan de inclusiecriteria in aanmerking, mits er geen sprake is van exclusiecriteria. Patiënten worden zowel tijdens kantooruren als tijdens ANW uren geïncludeerd, gezien het verschil in organisatie van huisartsenzorg tijdens kantooruren (eigen huisartspraktijk) en in ANW uren (huisartsenpost).

#### Inclusie- en exclusiecriteria

#### Inclusie:

- Patiënten van 18 jaar of ouder
- Patiënt wordt behandeld op de SEH gedurende inclusieperiode
- Patiënt is wilsbekwaam en heeft schriftelijk informed consent gegeven (indien patiënt geen toestemming kan geven kan de wettelijke vertegenwoordiger dit doen).
- Indien patiënt (of vertegenwoordiger) bij binnenkomst op de SEH niet in staat is informed consent te geven, kan dit door de hoofdonderzoeker alsnog binnen 24 uur na presentatie alsnog worden gevraagd.
- Hoofdbehandelaar is akkoord met inclusie

## Exclusie:

Taalbarrière

## Aantal beoogde proefpersonen

Het beoogde aantal proefpersonen is 750. Dit is een voldoende grote groep om uitspraken te kunnen doen over de patiënt journey binnen de acute zorgketen. Een sample size berekening is bij dit onderzoek niet van toepassing, mede gezien het exploratieve karakter van de studie.

## 2.3 Dataverzameling

## Methode

Van alle patiënten op de SEH worden basale gegevens verzameld (leeftijd, geslacht, urgentieclassificatie en verwezen specialisme). Na toestemming van de patiënt zullen overige gegevens verzameld worden middels een vragenlijst aan de patiënt (bijlage 1) en door raadpleging van het dossier van de patiënt (bijlage 2), inclusief de verwijsbrief van de huisarts. In de vragenlijst wordt gevraagd naar algemene patiënt karakteristieken en informatie over het verloop van de acute zorgketen. Het is te verwachten dat de onderzoeker samen met de patiënt en eventuele naasten de vragenlijst invult. Daarnaast wordt het dossier geraadpleegd door de onderzoeker om diverse gegevens te achterhalen en aan te vullen. Zo nodig kan de onderzoeker telefonisch bij de huisarts de ontbrekende data achterhalen. De zorg die patiënten ontvangen wordt niet door dit onderzoek beïnvloed. De vragenlijsten zullen mondeling en/of schriftelijk afgenomen worden, waarna ze direct in een database ingevoerd worden.

De betreffende hoofdbehandelaar zal op voorhand toestemming gevraagd worden voor het benaderen van zijn/haar patiënten.

Data zullen online opgeslagen worden in een elektronisch Case Report Form (eCRF), gemaakt met de Data Management module van Research Manager. Digitale data zal geanonimiseerd worden en gelabeld met een uniek nummer. De

coderingslijst, waarin deze gegevens zichtbaar zijn, zal op een separate locatie op de Zuyderland server, beveiligd met een wachtwoord, bewaard worden.

#### Verzamelen van data

Meerdere onderzoekers op diverse locaties. Coördinerend onderzoeker is drs. L. Claassen .

#### Standaardisering

De vragenlijst in bijlage 1 wordt voor iedere patiënt gebruikt.

## 2.4 Data-analyse

#### **Data-inspectie**

Missende waarden zullen zoveel mogelijk achterhaald worden via het dossier van de patiënt, verwijsinformatie die is overgedragen aan de SEH of door contact op te nemen met betrokken hulpverleners in de acute zorgketen. De data zullen steekproefsgewijs gecontroleerd worden door een tweede onderzoeker. De database wordt gecontroleerd op outliers of onwaarschijnlijke waarden en zo nodig gecontroleerd en gecorrigeerd worden.

## **Testen normale verdeling**

Visueel en middels Kolmogorov-Smirnov en de voor normaliteit specifieke Shapiro-Wilk-toets

## Beschrijvende statistiek

Alle data zal middels IBM SPSS statistische software 26 en Graphpad Prism 8 worden geanalyseerd. Beschrijvende statistiek zal worden toegepast op de verzamelde data middels de vragenlijsten en verwijsbrieven van de huisartsen om een inzicht te geven op de onderzoeksvraag naar de patient journey binnen de acute zorgketen van volwassen patiënten die behandelt worden op een SEH. Normaal verdeelde data zullen weergegeven worden als gemiddelden met standaarddeviatie, niet normaal verdeelde data als mediaan met interquartile range (IQR) en vergeleken met de Student T toets en Mann-Whitney U test, resp.. Categorische data wordt als absolute getallen weergegeven en percentages van subgroepen (leeftijd, ziekte, etc.) zal worden vergeleken met de chi-kwadraat test of de Fisher-exact test. Patronen in duur of samenstelling van prehospitale periode zullen tevens grafisch weergegeven worden, bijvoorbeeld om de associatie van leeftijd in het proces, de urgentie, de onderzoeken die op de SEH plaatsvinden etc. te onderzoeken.

#### **Codering en interpreteren**

De open antwoorden op alle vragen uit de vragenlijst zullen door het voltallige onderzoeksteam bekeken worden en worden gecategoriseerd. Deze informatie zal gebruikt worden om eventuele toekomstige studies te optimaliseren.

## Softwareprogramma

**IBM SPSS 26** 

## 2.5 Datamanagement

## Locatie

Data zullen online opgeslagen worden in een elektronisch Case Report Form (eCRF), gemaakt met de Data Management module van Research Manager. Digitale data zal geanonimiseerd worden en gelabeld met een uniek nummer. De coderingslijst, waarin deze gegevens zichtbaar zijn, zal op een separate locatie op de Zuyderland server, beveiligd met een wachtwoord, bewaard worden.

## **Toegang**

Alle leden van het onderzoeksteam hebben toegang tot de onderzoeksgegevens.

#### Bewaren van gegevens

15 jaar

## Beveiliging van gegevens

De database is enkel toegankelijk met een wachtwoord, welke persoonsgebonden is. Ook de coderingslijst is met een wachtwoord beveiligd. Data wordt opgeslagen op een beveiligde locatie.

#### Inzage patiëntendossier

Er worden voor deze studie alleen gegevens uit het patiëntendossier gehaald die relevant zijn voor de onderzoeksvraag en nadat toestemming is verkregen van de patiënt middels het informed consent formulier. De (werk)diagnose bij ontslag van SEH wordt door de onderzoeker genoteerd na overleg met de hoofdbehandelaar.

#### Codering

Data worden ingevoerd door de onderzoeker. Na toekenning van een uniek nummer aan de digitale data, zullen naam, geslacht, geboortedatum en patiëntnummer in een separate coderingslijst opgeslagen worden. Dit document wordt beveiligd met een wachtwoord op de Zuyderland server opgeslagen.

#### Codesleutel

Enkel de hoofdonderzoeker heeft na inclusie van de patiënten toegang tot de codesleutel.

#### Bescherming van privacy

Data worden gecodeerd opgeslagen in een eCRF, vanwaar uit de onderzoeksdatabase gecreëerd wordt. Deze data staan op een beveiligde server van Zuyderland. Op een separate locatie staat de coderingslijst, welke eveneens met een wachtwoord beveiligd wordt.

## Delen van gegevens

De gegevens worden alleen met betrokken onderzoekers op locaties buiten het Zuyderland gedeeld.

## **3 ETHISCHE OVERWEGINGEN**

## 3.1 Verklaring akkoord niet-WMO

Dit protocol zal worden ingediend bij METC-Z.

## 3.2 Belasting, risico en vergoeding voor proefpersonen

De belasting van de proefpersoon bestaat uit het beantwoorden van de vragen genoemd in bijlage 1. Dit duurt hooguit enkele minuten. Er is geen risico verbonden aan deelname aan de studie.

Indien een patiënt in verband met ernst van ziekte niet bij binnenkomst geïncludeerd kan worden, kan binnen 24u alsnog inclusie plaatsvinden door de onderzoeker.

## 3.3 Toestemming proefpersoon

| ois resistanting proceptions | |
|---|---|
| Prospectief niet-WMO | niet-WMO plichtig onderzoek: Informed Consent procedure |
| Benadering | De patiënt wordt op de SEH benaderd door onderzoeker, een A(N)IOS, een SEH-arts <sup>KNMG</sup> of |
| proefpersonen | medisch specialist en gevraagd of hij/zij wil deelnemen aan de studie. |
| Informeren | Aan iedere potentiële proefpersoon wordt mondeling en schriftelijk informatie verstrekt. |
| proefpersonen | Bij vragen kunnen deze aan de onderzoeker, de A(N)IOS, de SEH-arts <sup>KNMG</sup> of medisch specialist gesteld worden. |
| Bedenktijd | De proefpersoon kan op de SEH besluiten al dan niet mee te doen. Gezien de lage belasting en de afwezigheid van risico voor de patiënt lijkt het ons niet noodzakelijk een langere bedenktijd in te voeren. Tevens kan er dan de mogelijkheid tot recall bias ontstaan welke invloed kan hebben op de studieresultaten. Patiënten mogen uiteraard alsnog hun toestemming terugtrekken, data worden dan verwijderd. |
| Tekenen<br>toestemmings-<br>verklaring | De toestemmingsverklaring wordt op de SEH getekend. Deze toestemming is alleen noodzakelijk voor patiënten die benaderd worden door de onderzoekers en de vragenlijsten op de SEH invullen en het dossier van wordt ingezien. Van de patiënten die niet geïncludeerd worden (geen toestemming of gemist) zullen alleen de basale kenmerken (leeftijd, geslacht, urgentieclassificatie op de SEH en verwezen specialisme) worden verzameld, daar dit retrospectief verzamelde data is en naar verwachting > 50 personen omvat, is hier geen separate toestemming voor genoodzaakt. |

## **4 VALORISATIE EN PUBLICATIE**

## **Valorisatie**

De resultaten van dit onderzoek zullen gebruikt worden om gericht vervolgonderzoek op te zetten naar de patient journey door en organisatie van de acute zorgketen bij patiënten die uiteindelijk op de SEH behandeld worden met als doel verbeterplannen te maken voor het huidige acute zorglandschap. Specifiek gaat het om mogelijke punten binnen de zorgketen waar onnodige of vermijdbare vertraging optreedt.

#### **Publicatie**

De resultaten van dit onderzoek zullen aangeboden worden ter publicatie in een internationaal wetenschappelijk tijdschrift. Daarnaast worden ze tenminste regionaal besproken binnen het Netwerk Acute Zorg Limburg (NAZL).

## **REFERENTIES**

- 1 Latten GHP, Claassen L, Jonk M, et al. Characteristics of the prehospital phase of adult emergency department patients with an infection: A prospective pilot study. *PLoS One* 2019;14:e0212181 doi:10.1371/journal.pone.0212181 [doi].
- $2\ https://www.volksgezondheidenzorg.info/onderwerp/acute-zorg/cijfers-context/gebruik-acute-zorg\#node-gebruik-seh-naar-diagnose$
- 3 Westert G, Jabaaij L, Schellevis FG, eds. Morbidity, Performance and Quality in Primary Care. Dutch general practice on stage. Abingdon: Radcliffe Publishing Ltd 2006.
- 4 Stassen PM, Cals JW. Flashmobstudies: wetenschap in een flits. Ned Tijdschr Geneeskd 11 mei 2020;164:D4736.

| BIJLAGEN |
|--------------|
| BULAGEN |
| D.027 (G2.1) |

| Patient#: |
|------------------|
| Inclusielocatie: |

## Bijlage 1 – vragenlijst patiënt TACC studie – Time within the Acute Care Chain

Geachte heer/mevrouw,

ALGEMEEN

Graag willen we meer weten over wat er gebeurd is vanaf het moment dat u ziek werd totdat u nu bij ons op de spoedeisende hulp (SEH) gekomen bent. Dit willen we graag doen door middel van een aantal vragen, die u slechts enkele minuten van uw tijd zullen kosten. Wij danken u bij voorbaat voor deelname aan dit onderzoek.

 $\bigcirc$  Man

| 1. | desiaciit | ○ Vrouw |
|---|---|---|
| 2. | Leeftijd | jaar |
| 3. | Opleidingsniveau | <ul><li>Geen opleiding</li></ul> |
| vóó | R UW BEZOEK AAN DE SPOEDEISENDE HULP (SEH) <u>VANDAAG</u> | |
| 4. | Sinds welke datum heeft u deze klachten waarvoor u <u>nu</u> op de Spoedeisende hulp bent? | |
| 5. | Heeft u de afgelopen dagen naast het contact waarmee u op<br>de spoedeisende hulp bent gekomen (dus het contact van<br>vandaag niet meegeteld), eerder contact gehad met een<br>zorgverlener (huisarts, ambulance, medische hulplijn, dokter<br>in het ziekenhuis) | ◯ Ja<br>◯ Nee |
| 6. | Wanneer was het eerste contact met een zorgverlener in deze ziekte periode? | |
| 7. | Hoe vaak heeft u sinds uw eerste contact genoemd bij vraag 6, contact gehad met een zorgverlener (huisarts, ambulance, medische hulplijn, dokter in het ziekenhuis)? | keer, inclusief het eerste contact en het contact van vandaag |

| 8. | Werd er al medicatie aan u voorgeschreven? | <ul><li>○ Nee</li><li>○ Ja,</li><li>Datum:</li></ul> |
|---|---|---|
| 9. | Welke medicatie werd er voorgeschreven? | |
| UW E | BEZOEK AAN DE SPOEDEISENDE HULP (SEH) <u>VANDAAG</u> | |
| 10. | Met welke klacht of symptomen komt u vandaag? | |
| 11. | Door wie bent u vandaag verwezen? | <ul><li>Huisarts</li><li>Verpleeghuisarts</li><li>Medewerker ziekenhuis</li><li>Ambulance</li><li>Anders, nl</li></ul> |
| 12. | Hoe laat heeft u vandaag de verwezen zorgverlener gecontacteerd? | Tijdstip: uur Nee, ik heb eerder contact gehad maar ik kon pas vandaag terecht |
| 13. | Hoe laat hebt u de huisarts vandaag bezocht, of kwam deze bij u thuis? | Tijdstip: uur |
| 14. | Bent u vandaag met de ambulance naar de SEH gekomen? | ○ Ja<br>○ Nee; |
| 15. | Welke diagnose is er uiteindelijk door de dokter op de SEH gesteld? | |

# Bijlage 2 – vragenlijst patiënt TACC studie – Time within the Acute Care Chain

| Patient#: |
|------------------|
| Inclusielocatie: |

Vragenlijst door onderzoeker in te vullen met gegevens patiënten dossier.

| | ALGEMEEN | |
|---|---|---|
| 1. | Verwezen specialisme | |
| 2. | Verwezen door | <ul> <li>Huisarts, ga naar vraag 3</li> <li>Verpleeghuisarts</li> <li>Medewerker ziekenhuis</li> <li>Ambulance, ga naar vraag 4</li> <li>Anders, nl</li> </ul> |
| 3. | Klacht bij aanmelden | |
| 4. | Indien patiënt via HAP verwezen, wat was het urgentieniveau? | |
| 5. | Tijdstip aankomst ambulance bij patiënt | Tijdstip:: uur |
| 6. | Urgentieniveau van ambulance | |
| 7. | Datum + tijdstip ten tijde van <u>binnenkomst</u> op SEH | <br>Tijdstip:: uur |
| 8. | Urgentieniveau op SEH | |
| 9. | Datum + tijdstip ten tijde van <u>verlaten</u> op SEH | <br>Tijdstip:: uur |
| 10. | Diagnose bij verlaten SEH | |
| 11. | Welke onderzoeken zijn verricht tijdens het verblijf op de<br>SEH? (In te vullen door onderzoeker) | <ul> <li>○ Bloedonderzoek</li> <li>○ ECG</li> <li>○ Röntgenfoto</li> <li>○ Echografie</li> <li>○ CT-scan</li> <li>○ Anders, nl</li> </ul> |
| 12. | Wat is er gebeurd na de SEH? | Opname, ga naar vraag 12 Naar huis, ga naar vraag 14 ELV bed Anders, nl |
| 13. | Op welke afdeling werd patiënt opgenomen? | <ul><li>Gewone verpleegafdeling</li><li>High care afdeling zoals een MC, Hartbewaking of Brain Care</li><li>IC</li></ul> |
| 14. | Ontslagdatum | |

| 15. | Is patiënt nog in leven 7 dagen na presentatie op de SEH? | <ul><li>○ Ja</li><li>○ Nee, ga naar vraag 17</li></ul> |
|---|---|---|
| 16. | Is patiënt nog in leven 30 dagen na presentatie op de SEH? | <ul><li>○ Ja</li><li>○ Nee, ga naar vraag 17</li></ul> |
| 17. | Datum van overlijden | |
| 18. | Heeft de patiënt de SEH nogmaals bezocht? | <ul><li>○ Ja, ga naar vraag 19</li><li>○ Nee</li></ul> |
| 19. | Hoe vaak heeft de patiënt de SEH nogmaals bezocht na eerste presentatie? | keer |